CLINICAL TRIAL: NCT01024946
Title: Phase II Study of Everolimus (RAD001) for the Treatment of Malignant Pleural Mesothelioma With Merlin/NF2 Loss as a Biomarker to Predict Sensitivity
Brief Title: Everolimus (RAD001) for the Treatment of Malignant Pleural Mesothelioma With Merlin/NF2 Loss as a Biomarker to Predict Sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Dana-Farber Cancer Institute (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-142
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: mesothelioma; pleural; RAD001; Everolimus; 09-142; thoracic; lung; epithelioid; sarcomatoid
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Everolimus

ARMS (1):
- Pts getting everolimus (Experimental): This is a multicenter, open label, phase II study of everolimus as a second or third line therapy for the treatment of advanced malignant pleural mesothelioma, which will also evaluate Merlin/NF2 loss as a biomarker to predict sensitivity to everolimus. Patients who have disease progression after one or two prior chemotherapy regimens will be eligible. In the first stage of this design, 19 patients will be accrued. If 6 or less patients among the first 19 patients show clinical benefit, then the study will be terminated and declared negative. If 7 or more patients show clinical benefit, than an additional 20 patients will be accrued to the second stage. At the end of the study, if 17 or more patients show clinical benefit out of a total of 39 patients enrolled, the regimen will be considered worthy of further investigation.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — Everolimus will be administered at a dose of 10mg orally once daily continuously. Dose reduction may be required depending on the type and severity of toxicity encountered. One cycle will be considered 28 days. Patients will have CT scans to evaluate for response after cycle 1 and cycle 2, and then every two cycles thereafter.

SUMMARY:
For patients with malignant pleural mesothelioma that has grown despite treatment with standard chemotherapy, no treatment has yet proven beneficial. The purpose of this study is to find out what effects, both good and bad, that everolimus has on the cancer. Everolimus works by blocking a protein that helps the cancer grow. The goal of this clinical research study is to learn if the study drug everolimus can shrink or slow the growth of mesothelioma. The safety of this drug will also be studied. The patients' physical state, changes in the size of the tumor, and laboratory findings taken during the study will help us decide if everolimus is safe and effective.

DETAILED DESCRIPTION:
This is a multicenter, open label, phase II study of everolimus as a second or third line therapy for the treatment of advanced malignant pleural mesothelioma, which will also evaluate Merlin/NF2 loss as a biomarker to predict sensitivity to everolimus. Patients who have disease progression after one or two prior chemotherapy regimens will be eligible. In the first stage of this design, 19 patients will be accrued. If 6 or less patients among the first 19 patients show clinical benefit, then the study will be terminated and declared negative. If 7 or more patients show clinical benefit, than an additional 20 patients will be accrued to the second stage. At the end of the study, if 17 or more patients show clinical benefit out of a total of 39 patients enrolled, the regimen will be considered worthy of further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of epithelioid, sarcomatoid, or mixed-type malignant pleural or peritoneal mesothelioma that is not amenable to surgery.
* Patients must have measurable disease according to the modified RECIST criteria for mesothelioma.
* Patients must have adequate tissue sample available for analysis of NF2/Merlin loss. (archived tissue block or 10 unstained slides)
* Patients must have received no more than two prior systemic therapy regimens, and at least one of the regimens must have included pemetrexed.
* Patients must be at least 18 years of age.
* Karnofsky performance status > or = to 70%.
* Adequate renal function: serum creatinine ≤ 1.5 x ULN.
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent
* Patients must have adequate hepatic function as defined by:

  * AST and ALT ≤ 2.5 x ULN (≤ 5x ULN in patients with liver metastases)
  * Serum bilirubin ≤ 1.5 x ULN
* Patients must have adequate bone marrow function as defined by:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL

Exclusion Criteria:

* Patient has been previously treated with an mTOR inhibitor (sirolimus, temsirolimus, or everolimus).
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 3 weeks of the start of study drug for chemotherapy, biologics, targeted therapies, or immunologics or 2 weeks for radiation provided that patients have recovered from all associated toxicities at the time of registration
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids (except with a dosage equivalent to ≤ prednisone 20 mg) or another immunosuppressive agent. Patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first planned treatment with everolimus. Topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one week of study entry.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * uncontrolled diabetes as defined by fasting serum glucose > or = to 1.5 x ULN
* Severely impaired lung function as evidenced by:

  o DLCO < 35% of the normal predicted value and/or O2 saturation that is ≤ 88% at rest on room air
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus)
* Patient has an active infection for which they received IV antibiotic, antiviral, or antifungal medications within 2 weeks of starting study drug.
* Patients with a "currently active" second malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Krug, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Getting Everolimus: This is a multicenter, open label, phase II study of everolimus as a second or third line therapy for the treatment of advanced malignant pleural mesothelioma, which will also evaluate Merlin/NF2 loss as a biomarker to predict sensitivity to everolimus. Patients who have disease progression after one or two prior chemotherapy regimens will be eligible. In the first stage of this design, 19 patients will be accrued. If 6 or less patients among the first 19 patients show clinical benefit, then the study will be terminated and declared negative. If 7 or more patients show clinical benefit, than an additional 20 patients will be accrued to the second stage. At the end of the study, if 17 or more patients show clinical benefit out of a total of 39 patients enrolled, the regimen will be considered worthy of further investigation.
  everolimus: Everolimus will be administered at a dose of 10mg orally once daily continuously. Dose reduction may be required depending on the type and severity
Period: Overall Study
Arm/Group | Patients Getting Everolimus
Started | 11
Completed | 6
Not Completed | 5
Not completed — Screen Failure | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Getting Everolimus
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Rate of Clinical Benefit (i.e. Rate of Complete or Partial Response Plus Stable Disease) at 16 Weeks for Patients With Malignant Mesothelioma Treated With Everolimus as Second or Third Line Therapy.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Patients Getting Everolimus
Number analyzed (Participants) | 6
participants
  Stable Disease | 4
  Progression of Disease | 2

ADVERSE EVENTS:
Arm/Group | Patients Getting Everolimus
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Getting Everolimus (N=7)
Constipation (Gastrointestinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inf norm ANC/gr1/2 neut-Myositis infection(muscle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 (1)
Ascites (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Getting Everolimus (N=7)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4)
ALT, SGPT (Metabolism and nutrition disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (6)
Glucose, high (hyperglycemia) (Blood and lymphatic system disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes